CLINICAL TRIAL: NCT04630691
Title: Evaluation of Posterior Narrow Diameter Implants in Hyperglycemic and Normo-glycemic Patients
Brief Title: Posterior Narrow Diameter Implants in Hyperglycemic and Normo-glycemic Patients
Status: Completed | Type: Observational
Sponsor: University of Witten/Herdecke (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Other Study IDs: UWHPerioT2DM
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2; Implant Complication
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Drug Implants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Patients with HbA1c around 6,0
  Interventions: Procedure: Implantation
- T2DM: Patients with HbA1c above 6,5
  Interventions: Procedure: Implantation

INTERVENTIONS:
Procedure: Implantation — Patients received narrow diameter implants in posterior mandible or maxilla

SUMMARY:
The aim of the present study was to compare the initial healing and long term performance of narrow diameter implants in patients with uncontrolled Diabetes mellitus type 2 (T2DM) and healthy individuals.

ELIGIBILITY:
Inclusion criteria:

Patients with one or more missing teeth posterior to the canine either in the maxilla or mandible and associated with diminished alveolar ridge dimensions were included in the study

Exclusion Criteria:

* immobility of diabetic patients
* periodontal surgery and/or antibiotic therapy within the last 6 months prior to baseline
* pregnancy and lactation period
* Full Mouth Plaque Score (FMPS) > 25%
* untreated periodontitis
* smoking > 10 cigarettes/day
* insufficient crestal volume making an augmentation procedure necessary
* previously performed ridge augmentation procedure for a staged implant placement
* permanent medication potentially affecting blood perfusion rate and bone metabolism

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
No difference | 3 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diehl D, Bespalov A, Yildiz MS, Friedmann A. Restoration of posterior teeth by narrow diameter implants in hyperglycemic and normoglycemic patients - 4-year results of a case-control study. Clin Oral Investig. 2024 Jun 22;28(7):392. doi: 10.1007/s00784-024-05786-0. PMID 38907052
- [Derived] Diehl D, Kaner D, Bockholt A, Bilhan H, Friedmann A. Microcirculation and neutrophil-related cytokine concentrations are not altered around narrow diameter implants in T2DM patients during wound healing. Clin Oral Investig. 2023 Mar;27(3):1167-1175. doi: 10.1007/s00784-022-04731-3. Epub 2022 Oct 13. PMID 36229741
- [Derived] Friedmann A, Winkler M, Diehl D, Yildiz MS, Bilhan H. One-year performance of posterior narrow diameter implants in hyperglycemic and normo-glycemic patients-a pilot study. Clin Oral Investig. 2021 Dec;25(12):6707-6715. doi: 10.1007/s00784-021-03957-x. Epub 2021 May 3. PMID 33939006